CLINICAL TRIAL: NCT01750164
Title: Patient Derived Breast Cancer Xenografts
Status: Terminated | Type: Observational
Why Stopped: discontinued funding
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D12168
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2013-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and tumor tissue samples as well as DNA that has been extracted from both blood and tiisue will be stored.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Invasive breast cancer with metastatic disease

SUMMARY:
This study will use tissue or body fluid acquired during standard procedures that are part of the patient's care for their cancer, such as surgery to remove tumor tissue or needle withdrawal of body fluid containing cancer cells. The tissue or cells will be injected into immune compromised mice and the tissue will be allowed to grow to a tumor 1-1.5 cm size. The tissue will then be extracted and either frozen, embedded in paraffin, or used for engraftment into another generation of mice. The second generation mice will be separated into groups and given various treatments.

Tissue from the participants and from the mouse established tumors, in which the mice have either received treatment or have not received treatment, will be used to evaluate the levels of various genes that assist in regulating cell growth and cell death. The tumor tissue from participants and mice will also be tested for random changes in the genetic material and compared to the participant's blood to determine if any of the changes in the genetic material correlate with better engraftment of the patient tissue in the mice. It is anticipated that 10-30% will have successful engraftment of tumor tissue

ELIGIBILITY:
* Women > age 18. with a history of ER+. HER-2 negative breast cancer previously treated with adjuvant anti-estrogen therapy (tamoxifen or aromatase inhibitor? for at least 1 year after surgical resection of primary tumor.
* ER+ status requires positive staining in > 10% of malignant cells in biopsy specimen.
* HER-2 Negative status requires Immunohistochemistry 0-1+, or with a FISH ratio of < 2.0 if IHC is 2+ or if IHC has not been done.
* Patient must have: A. newly diagnosed recurrent, locally advanced or metastatic breast cancer. B. existing advanced or metastatic breast cancer.
* Patient must be having clinically indicated: A. diagnostic tumor biopsy via core-or needle incision or B. surgical removal of tumor or C. collection of pleural or ascetic fluid in order to obtain fresh tumor tissue for research (transplant into mice).
* For subjects having a diagnostic tumor biopsy, excess fresh tumor tissue must be available from the biopsy for research for immediate transplantation into mice.
* For subjects having a surgical resection of the primary tumor, the tumor must have a clinical size of 1 cm or greater, and and excess fresh tumor tissue must be available from the surgical specimen for research for immediate transplantation into mice.
* Ability to give signed informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with invasive breast cancer with metastatic disease seen in Oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Successful Engraftment | 2 years
  Thirty-five patients with breast cancer will be recruited. We anticipate that 10-30% will have successful engraftment of tumor tissue. The achievement of five successful xenografts would justify additional study.

SECONDARY OUTCOMES:
Time until tumor formation | 2 years
  The rate of tumor growth will be calculated. Mice are monitored three times per week for general health and tumor length. Tumor length Tumor length and width are measured with calipers and recorded. Tumor volume will be calculated with the formula (Length x Width x Width)/2, derived from the formula for the volume of an ellipsoid. Tumor growth will be measured at each time point by calculating the ratio of tumor volume (V) to the initial tumor volume (Vo). Average time, measured in weeks, required for tumors to form palpable masses in F1 mice will be recorded as the Time-until-Tumor-Formation (TTF). A comparison of TTF between tumor cells isolated from tumor tissue isolated by surgical biopsy, and by malignant cells in a body fluid will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Gary Schwartz, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States